CLINICAL TRIAL: NCT05001828
Title: Phase IA/B Combination Study of ADI-PEG 20, Venetoclax and Azacitidine in Patients With Acute Myeloid Leukemia (AML)
Brief Title: Study of ADI-PEG 20, Venetoclax and Azacitidine in Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2020-002
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ADI PEG20; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Previously Treated AML (Experimental): Previously treated AML based on the revised revised 2022 WHO criteria with age at least 18 years.
  Interventions: Drug: ADI-PEG 20
- Untreated AML With High Risk Features (Experimental): Untreated AML per 2022 WHO criteria with high-risk features and not a candidate for intensive chemotherapy because of age 60 years or older, age-related comorbidities, cardiac disease, prior anthracycline use, high probability of treatment-related mortality, or otherwise would not benefit from intensive chemotherapy treatment.
  Interventions: Drug: ADI-PEG 20

INTERVENTIONS:
Drug: ADI-PEG 20 — ADI-PEG 20 in combination with venetoclax and azacitidine
  Other Names: Venetoclax; Azacitidine

SUMMARY:
Pegylated arginine deiminase (ADI-PEG 20) will be combined with venetoclax and azacitidine for treatment of subjects with previously treated or untreated with high risk factor acute myeloid leukemia (AML). Venetoclax and azacitidine are front-line therapy for such patients, and ADI-PEG 20 will be added to this regimen in a phase IA/B study.

DETAILED DESCRIPTION:
This is an open label, single arm, phase 1 trial with recommended phase 2 dose (RP2D) cohorts based on subject inclusion criteria.

Lead In: 6 patients will be enrolled to be treated with standard dose of azacitidine and venetoclax and the expected RP2D of ADI-PEG 20 (dose level 0). In case of DLT occurring in >1 patient in cycle 1, 6 additional patients will be accrued at dose level -1 of ADI-PEG 20 while keeping the doses of azacitidine and venetoclax unchanged (Dose level -1). Enrollment to cohort 1 and 2 will start after ≤1 patient out of 6 encounters DLT in cycle 1 at one of these dose levels. The 6 patients enrolled at that dose level will be counted for efficacy analysis. Cohort 1: Relapsed or refractory AML: target response 25%. Historical expectation for venetoclax and azacitidine is 15%.

Cohort 2: Newly diagnosed high risk AML: Target response 55%. Historical expectation for venetoclax and azacitidine is 40%.

Treatment may be continued for a maximum of 24 cycles or 104 doses of ADI-PEG 20 (study Week 103), whichever is reached first.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Previously treated (relapsed/recurrent) or refractory AML based on the 2022 revision to the World Health Organization (WHO) criteria (Arber 2022)
* Cohort 2: Untreated AML per 2022 WHO (Arber 2022) criteria with high-risk features and not a candidate for intensive chemotherapy because of age 60 years or older, age-related comorbidities, cardiac disease, prior anthracycline use, high probability of treatment-related mortality, or otherwise would not benefit from intensive chemotherapy treatment.
* Age ≥ 18 years
* Life expectancy reasonably adequate for evaluating the treatment
* White blood cell (WBC) count of 10 × 109/L or less. (Use of hydroxyurea to control WBC is allowed till 48 hours prior to protocol treatment)
* Adequate renal function: Creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance > 40 mL/minute (measured or calculated according to the Cockcroft-Gault formula)
* Adequate liver function

  * Total bilirubin ≤ 1.5 x ULN
  * ALT and AST both ≤ 2.5 x institutional ULN or ≤ 5 times the ULN for patients with leukemic involvement of liver

Exclusion Criteria:

* Prior treatments as follows:

  1. Cohort 1: >2 cycles of prior combination treatment with venetoclax+hypomethelating agent (i.e. azacitidine, decitabine) is exclusionary. All other prior treatment for antecedent hematological disorders and/or for AML is permitted.
  2. Cohort 2: Prior treatment for antecedent hematological disorders with venetoclax or chemotherapy or any prior treatment for their AML is exclusionary. However, treatment with other agents, including hydroxyurea or ≤2 cycles of hypomethylating agent (i.e. azacitidine, decitabine), for MDS or myeloproliferative neoplasm is permitted.
* Cohort 2: Favorable risk AML per European LeukemiaNet (ELN) 2022 criteria (Döhner 2022)
* Known active CNS involvement by leukemia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine the RP2D of ADI-PEG 20 in combination with venetoclax and azacitidine, per the number of subjects with treatment-related adverse events by current CTCAE | 6 months

SECONDARY OUTCOMES:
Determine preliminary evidence of tumor activity, per the revised 2017 European LeukemiaNet criteria | 2 years
Determine the peripheral blood arginine levels of ADI-PEG 20 in combination with venetoclax and azacitidine | 2 years
Determine the peripheral blood citrulline levels of ADI-PEG 20 in combination with venetoclax and azacitidine | 2 years
Determine the anti-drug antibodies of ADI-PEG 20 in combination with venetoclax and azacitidine | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John S Bomalaski, MD, Study Director — Polaris Group
Locations (3):
- United States (3):
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Levine Cancer Institute, Charlotte, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No